CLINICAL TRIAL: NCT00490919
Title: Multi-center, Randomized, Double-blind, Placebo-controlled With Open Label run-in Study Assessing Efficacy, Tolerability, Safety of BTDS 10 or 20 Compared to Placebo in Opioid-naïve Subjects With Moderate to Severe, Chronic Low Back Pain
Brief Title: Buprenorphine Transdermal System (BTDS) in Subjects With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3024
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Low Back Pain
Keywords: Chronic pain; opioid; transdermal; Moderate to severe chronic low back pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double-blind BTDS 10 or 20 (Experimental): Buprenorphine transdermal system 10 or 20 mcg/h applied for 7-day wear
  Interventions: Drug: Buprenorphine transdermal system
- Double-blind Placebo TDS (Placebo Comparator): Placebo transdermal system to match BTDS patches, applied for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine transdermal system — Buprenorphine transdermal system 10 or 20 mcg/h worn for 7 days
  Other Names: Butrans™
  Arms: Double-blind BTDS 10 or 20
Drug: Placebo — transdermal system (placebo) worn for 7 days
  Arms: Double-blind Placebo TDS

SUMMARY:
The objective of this study is to determine the analgesic efficacy and safety of Buprenorphine Transdermal System (BTDS) 10 and 20 compared to placebo in opioid-naïve subjects with moderate to severe chronic low back pain. The double-blind treatment intervention duration is 12 weeks, during which time supplemental analgesic medication (immediate-release oxycodone for the first 6 days post-randomization and acetaminophen or ibuprofen for the remainder of the double-blind phase) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic settings for the relief of moderate to severe pain. BTDS is a transdermal system formulation that is designed to deliver a consistent and a steady dose of buprenorphine over a 7-day period with limited blood concentration fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe chronic low back pain (lasting several hours daily) as their predominant pain condition for at least 3 months prior to screening,
* Subjects treated within the 14 days prior to screening with nonopioid therapy only, or with therapy including opioids at a dose of <5 mg oxycodone (or equivalent) per day,
* Subjects whose low back pain is not adequately controlled with non-opioid analgesic medication and who the Investigator feels are appropriate candidates for around-the-clock opioid therapy

Exclusion Criteria:

* Subjects who had a surgical procedure directed towards the source of back pain within 6 months of screening or planned during the study conduct period,
* Subjects who are allergic to buprenorphine or who had a history of allergies to other opioids,
* Subjects who have allergies or other contraindications to transdermal delivery systems or patch adhesives.

Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (79):
  - Research Facility, Anniston, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Radiant Research; Phoenix Southeast, Chandler, Arizona
  - Arizona Research Center Inc., Phoenix, Arizona
  - Research Facility, Phoenix, Arizona
  - Research Facility, Anaheim, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Research Facility, Carmichael, California
  - Advance Care Medical Group, City of Industry, California
  - Research Facility, Downey, California
  - Research Facility, Foothill Ranch, California
  - Research Facility, Sacramento, California
  - Research Facility, San Luis Obispo, California
  - Research Facility, Littleton, Colorado
  - Research Facility, Stamford, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Research Facility, Clearwater, Florida
  - University Clinical Research, DeLand, Florida
  - Arthritis Associates of S. FL, Delray Beach, Florida
  - Research Facility, Fort Myers, Florida
  - Century Clinical Research, Inc., Holly Hill, Florida
  - Research Facility, Jupiter, Florida
  - Research Facility, Largo, Florida
  - Research Facility, Merritt Island, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Plantation, Florida
  - Research Facility, Port Orange, Florida
  - Clinical Research of West Flor, Tampa, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, West Palm Beach, Florida
  - Independent Neurodiagnostic Clinic, Atlanta, Georgia
  - Research Facility, Dawsonville, Georgia
  - Druid Oaks Health Center, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Honolulu, Hawaii
  - Research Facility, Boise, Idaho
  - Rehabilitation Association of IN, Indianapolis, Indiana
  - Research Facility, Overland Park, Kansas
  - CTT Consultants, Inc., Prairie Village, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Research Facility, New Orleans, Louisiana
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Brockton, Massachusetts
  - East Coast Clinical Research, Haverhill, Massachusetts
  - Research Facility, Springfield, Massachusetts
  - Research Facility, Bay City, Michigan
  - Research Facility, Biloxi, Mississippi
  - Research Facility, Florissant, Missouri
  - Research Facility, St Louis, Missouri
  - Sports Med Consultants, PC, St Louis, Missouri
  - Research Facility, Henderson, Nevada
  - Research Facility, Las Vegas, Nevada
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Research Facility, New York, New York
  - Research Facility, Charlotte, North Carolina
  - Research Facility, Greensboro, North Carolina
  - Research Facility, Morgantown, North Carolina
  - Research Facility, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Research Facility, Columbus, Ohio
  - Research Facility, Toledo, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Eugene, Oregon
  - Research Facility, Medford, Oregon
  - Research Facility, Altoona, Pennsylvania
  - Research Facility, Chicora, Pennsylvania
  - Research Facility, Duncansville, Pennsylvania
  - Research Facility, Mechanicsburg, Pennsylvania
  - Research Facility, West Reading, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Anderson Family Care, PA, Anderson, South Carolina
  - KRK Medical Research, Dallas, Texas
  - Research Facility, Killeen, Texas
  - Research Facility, Plano, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Sugarland, Texas
  - Research Facility, Salt Lake City, Utah
  - Research Facility, Roanoke, Virginia

REFERENCES:
- [Result] Steiner DJ, Sitar S, Wen W, Sawyerr G, Munera C, Ripa SR, Landau C. Efficacy and safety of the seven-day buprenorphine transdermal system in opioid-naive patients with moderate to severe chronic low back pain: an enriched, randomized, double-blind, placebo-controlled study. J Pain Symptom Manage. 2011 Dec;42(6):903-17. doi: 10.1016/j.jpainsymman.2011.04.006. Epub 2011 Sep 25. PMID 21945130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study dates: 27-Jun-2007 (first patient first visit) to 24-Jul-2008 (last patient last visit), at 86 medical/research sites in the USA.
Pre-assignment Details: The open-label run-in period (N = 1024 started) was designed to select subjects for randomization in the double-blind phase who met both tolerability and responsiveness criteria for either BTDS 10 or 20 (an enriched design).
Groups:
- Open-label Run-in Period: The open-label run-in period (< 27 days) (N = 1024 started) was designed to select subjects for randomization who met both tolerability and responsiveness criteria for either BTDS 10 or 20 (an enriched design).
  Upon completion of the run-in period, 541 subjects were randomized and received treatment in the double-blind phase. Two subjects had no safety data after the randomization visit; therefore N = 539 for the randomized safety population.
- Double-blind BTDS 10 or 20: Buprenorphine transdermal patch (BTDS) 10 mcg/h or 20 mcg/h applied for 7-day wear during the 12-week double-blind phase.
- Double-blind Placebo TDS: Matching placebo transdermal patch (placebo TDS) 10 or 20 mcg/h applied for 7-day wear during the 12-week double-blind phase.
Period: Open-label Run-in Period
Arm/Group | Open-label Run-in Period | Double-blind BTDS 10 or 20 | Double-blind Placebo TDS
Started | 1024 | 0 | 0
Completed | 541 (Completed run-in and randomized; however 2 had no safety data after randomization visit (N = 539)) | 0 | 0
Not Completed | 483 | 0 | 0
Not completed — Adverse Event | 239 | 0 | 0
Not completed — Withdrawal by Subject | 37 | 0 | 0
Not completed — Lost to Follow-up | 21 | 0 | 0
Not completed — Lack of Efficacy | 143 | 0 | 0
Not completed — Administrative | 40 | 0 | 0
Not completed — Confirmed or suspected diversion | 3 | 0 | 0
Period: Double-blind Phase
Arm/Group | Open-label Run-in Period | Double-blind BTDS 10 or 20 | Double-blind Placebo TDS
Started | 0 | 256 (1 subject had no safety data in DB phase; therefore is excluded from randomized safety population.) | 283 (1 subject had no safety data in DB phase; therefore is excluded from randomized safety population.)
Completed | 0 | 170 | 199
Not Completed | 0 | 86 | 84
Not completed — Adverse Event | 0 | 40 | 20
Not completed — Withdrawal by Subject | 0 | 10 | 11
Not completed — Lost to Follow-up | 0 | 8 | 11
Not completed — Lack of Efficacy | 0 | 22 | 36
Not completed — Administrative | 0 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Double-blind BTDS: Buprenorphine transdermal patch 10 mcg/h or 20 mcg/h applied for 7-day wear during the 12-week double-blind phase
- Double-blind Placebo TDS: Matching placebo TDS 10 or 20 mcg/h applied for 7-day wear during the 12-week double-blind phase
- Total: Total of all reporting groups
Arm/Group | Double-blind BTDS | Double-blind Placebo TDS | Total
Number analyzed (Participants) | 256 | 283 | 539
Age Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.50) | 50.1 (13.31) | 49.5 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 163 | 296
  Male | 123 | 120 | 243

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Over the Last 24 Hours Scores at Week 12 of the Double-blind Phase.
Description: Pain was assessed on an 11-point numerical scale ranging from 0 = no pain to 10 = pain as bad as you can imagine.
Time Frame: Prerandomization phase consisted of a 6-10 day screening period and a <27 day open-label run-in period; and a 12-week double-blind phase.
Population: The full analysis population (FAP) (N = 541) [539] consisted of subjects who were randomized and received at least 1 dose of the double-blind study drug. (Two subjects did not have safety data.)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-blind BTDS | Double-blind Placebo TDS
Number analyzed (Participants) | 256 | 283
Units on a scale
  Screening | 7.24 (1.263) | 7.17 (1.223)
  Prerandomization | 2.57 (1.283) | 2.56 (1.207)
  Week 12 - Primary outcome | 3.83 (2.738) | 4.38 (2.690)
Statistical Analysis 1: Comparison: Double-blind BTDS vs Double-blind Placebo TDS; Missing average pain over the last 24 hours scores after treatment discontinuation were imputed using BOCF for adverse event-related withdrawals and LOCF for withdrawals due to other reasons; Test type: Superiority or Other; p = .0104, Mixed Models Analysis; Mixed effects general linear model with repeated measures; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.02 to -0.14], Standard Error of Mean 0.225 — Double-blind analysis (comparison between BTDS and placebo TDS) at week 12 of the double-blind phase

2. Secondary Outcome: The Mean Daily Number of Tablets of Nonopioid Supplemental Analgesic Medications Taken During Weeks 2 Through 12 of the Double-blind Phase
Description: Nonopioid supplemental analgesic tablets were sponsor-supplied acetaminophen or ibuprofen.
Time Frame: weeks 2-12
Population: Subjects in the full analysis population who took at least one dose of supplemental analgesic medication.
Measure: Mean (Standard Error); unit: tablets
Arm/Group | Double-blind BTDS | Double-blind Placebo TDS
Number analyzed (Participants) | 137 | 180
tablets | 0.620 (0.0658) | 0.743 (0.0574)
Statistical Analysis 1: Comparison: Double-blind BTDS vs Double-blind Placebo TDS; Test type: Superiority or Other; p = .1586, ANCOVA — To address the issue of multiplicity and control the family-wise error rate, a gate-keeping strategy and a stepwise approach (Holms methodology) were used to evaluate the statistical significance of the secondary efficacy analyses; Mean Difference (Final Values) = -0.124, 95% CI 2-sided [-0.296 to 0.048], Standard Error of Mean 0.0874 — Mean comparison from weeks 2-12 of the double-blind phase

3. Secondary Outcome: The Sleep Disturbance Subscale in the Medical Outcome Study (MOS) Sleep Scale at Weeks 4, 8, and 12 of the Double-blind Phase
Description: The MOS Sleep Scale consists of 12 individual items (4 sleep disturbance, 2 sleep adequacy, 1 quantity of and optimal sleep, 3 somnolence, 1 snoring, and 1 shortness of breath) and takes 5 to 10 minutes to complete. Question 1 is scored on a scale of 1 to 5 and Questions 2 to 12 are scored on a scale of 1 to 6. The Sleep Disturbance Subscale score is derived from the scores to Questions 1, 3, 7 and 8, and ranges from 0 to 100, where higher scores indicate greater sleep disturbance.
Time Frame: Weeks 4, 8, 12 of double-blind phase
Population: The full analysis population (FAP) (N = 541) consisted of subjects who were randomized and received at least 1 dose of the double-blind study drug. 2 subjects did not have safety data (N = 539).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double-blind BTDS | Double-blind Placebo TDS
Number analyzed (Participants) | 256 | 283
Units on a scale
  Week 4 | 32.84 (25.552) | 41.20 (26.813)
  Week 8 | 35.63 (26.276) | 39.87 (26.362)
  Week 12 | 34.97 (26.871) | 40.42 (26.675)
Statistical Analysis 1: Comparison: Double-blind BTDS vs Double-blind Placebo TDS; The primary comparison between groups was based on estimates and contrasts for the weeks 4, 8, and 12 mean values; Test type: Superiority or Other; p = .0062, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mixed effects general linear model with repeated measures; Mean Difference (Final Values) = -4.40, 95% CI 2-sided [-7.55 to -1.25], Standard Error of Mean 1.605 — Treatment comparison over Weeks 4, 8, and 12

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) that occurred after the signing of the informed consent up to end of study and 7 days after, discontinuation, or Serious AEs occurring up to 30 days following the last study visit were followed until the AE resolved or stabilized.
Description: AEs were obtained through spontaneous reports, subject interview, and subject diaries.
Groups:
- Double-blind BTDS 10, 20: Buprenorphine transdermal patch 10 mcg/h or 20 mcg/h applied for 7-day wear
- Double-blind Placebo TDS 10, 20: Matching placebo TDS 10 or 20 applied for 7-day wear
- Open-label Run-in Period, BTDS 5, 10, 20: Open-label BTDS 5, 10, 20 applied for 7-day wear
Arm/Group | Double-blind BTDS 10, 20 | Double-blind Placebo TDS 10, 20 | Open-label Run-in Period, BTDS 5, 10, 20
Serious Adverse Events (participants affected / at risk) | 3/256 | 2/283 | 4/1024
Other Adverse Events (participants affected / at risk) | 52/256 | 63/283 | 437/1024
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind BTDS 10, 20 (N=256) | Double-blind Placebo TDS 10, 20 (N=283) | Open-label Run-in Period, BTDS 5, 10, 20 (N=1024)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
Homicidal thoughts (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Systematic and nonsystematic assessments
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Drug abuser (Social circumstances) | 1 (1) | 0 (0) | 0 (0) — Systematic and nonsystematic assessments
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind BTDS 10, 20 (N=256) | Double-blind Placebo TDS 10, 20 (N=283) | Open-label Run-in Period, BTDS 5, 10, 20 (N=1024)
Nausea (Gastrointestinal disorders) | 32 | 31 | 240 — Systematic and nonsystematic assessments were used.
Vomiting (Gastrointestinal disorders) | 11 | 5 | 77 — Systematic and nonsystematic assessments were used.
Constipation (Gastrointestinal disorders) | 9 | 3 | 67 — Systematic and nonsystematic assessments were used.
Application site pruritus (General disorders) | 11 | 19 | 87 — Systematic and nonsystematic assessments were used.
Application site erythema (General disorders) | 9 | 14 | 32 — Systematic and nonsystematic assessments were used.
Application site rash (General disorders) | 12 | 7 | 18 — Systematic and nonsystematic assessments were used.
Dizziness (Nervous system disorders) | 10 | 3 | 102 — Systematic and nonsystematic assessments were used.
Somnolence (Nervous system disorders) | 4 | 6 | 84 — Systematic and nonsystematic assessments were used.
Headache (Nervous system disorders) | 14 | 14 | 100 — Systematic and nonsystematic assessments were used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days